Testing Legally Feasible Options Studies 2/3 NCT05604508 November 6, 2024

## **Study Protocol**

**Study objective.** The overall objective of this research is to experimentally evaluate legally viable approaches to reducing the impact of the POS retail environment on adolescent risk of using four classes of tobacco products: cigarettes, ENDS, smokeless tobacco, and LCCs. This study will be investigating regulations for four classes of tobacco products (cigarettes, e-cigarettes, smokeless tobacco, little cigars/cigarillos). Study 2 and study 3 (out of 3 studies), occurring concurrently, will examine whether changing the number and price content of posters on the outside doors at POS reduced adolescents' tobacco use risk. The study took place in the RAND StoreLab, a life-sized replica of a convenience store.

**Study design.** The experimental conditions that we will compare in this study are the RSL displaying a larger number of tobacco posters (16 posters total) versus the RSL with a smaller number of tobacco posters (8 posters total); and the RSL displaying tobacco posters with price discount information on them versus the RSL displaying tobacco posters with no price discount information on them.

**Methods.** The study was approved by the RAND Human Subjects Protection Committee. Young people were recruited from the community through standard advertising campaigns. Interested individuals completed a telephone screening to determine eligibility. Eligible individuals completed informed consent. Participants completed a baseline questionnaire that assessed demographics, tobacco product cognitions, smoking and tobacco use, and convenience store shopping habits. Participants were then randomized to one of the three experimental conditions. They were provided with a \$20 (fake) RSL gift card and asked to shop in the RSL for whatever they wanted, for as long as they wanted. They were asked to purchase at least one item and check-out and pay for the item(s) as they would in any convenience store. A confederate who was not involved in the consent or survey process served as the cashier. This cashier scanned the selected items for a total price, scanned the gift card, and bagged the items. Although no participants attempted to purchase tobacco from the RSL in this study, any such attempts would have been met by the cashier with a request for age identification and the purchase attempt would have been declined (i.e., because no participants were > 21 years old). After exiting the RSL, participants completed the dependent measures. They then: underwent a graduated debriefing; were asked to guess the study's purpose; and were told that they would be unable to retain the items they selected from the RSL. Participants then viewed a short tobacco media literacy video and received printed smoking prevention materials. Finally, they received compensation for participating.

## Statistical analysis plan

First, we evaluated whether randomization distributed pre-shopping baseline characteristics evenly across the experimental conditions. These univariable analyses used either t-tests or chi-squared tests to evaluate significance (depending on variable distribution). Next, we used logistic regression to evaluate the relationship between the experimental conditions and post-RSL shopping risk of using cigarettes; ENDS LCCs, and smokeless tobacco. Models adjusted for age, gender, race, socioeconomic status, lifetime tobacco use, and baseline tobacco use risk.